CLINICAL TRIAL: NCT03506074
Title: Flavor Perception in the Population of Campania Region, Italy
Brief Title: Flavor Test Results in General Population
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Paolo Emidio Macchia, Prof., Federico II University
Other Study IDs: PM0001/18
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Weight, Body; Smoking; Age Problem
Keywords: Obesity; Flavor
MeSH Terms: conditions — Body Weight; Smoking; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population: Adult volunteers (≥18 years of age) selected as part of a project to investigate the role of lifestyle in preventing chronic diseases supported by the Campus Salute association (www.campussalute.it).
  All volunteers performed the flavor test as described in Maione et al, Endocrine, 2016 (doi:10.1007/s12020-015-0690-y).
  Interventions: Diagnostic Test: Flavor test

INTERVENTIONS:
Diagnostic Test: Flavor test — The flavor test was developed, validated and patented (patent no. 0001426253 of the Italian Ministry for the Economic Development). It consists of a series of 20 aromatic extracts, corresponding to routine dietary use flavors for Italian people. At each administration, participants were invited to identify the aromatic by making a choice from 5 proposed items. A total of 21 aromatics (including one blank) were administered sequentially. The flavor score (FS) was calculated as the sum of correctly identified aromatics and ranged from 0 to 21.

SUMMARY:
Dietary choices are influenced by several factors, including physiological, social or genetic factors. Among these, flavor is the most important determinant modulating the preferences versus specific foods.

Flavor perception is the result from the sensory integration of taste and odor properties of food.

Aim of the present study was to assess flavor abilities in a large population using a validated perceptive test.

DETAILED DESCRIPTION:
This protocol investigates flavor perception using the flavor test, a specific test to assess the retro-nasal olfactory function.

A decrease in taste and smell abilities can result in loss of appetite, inadequate dietary intake and malnutrition. Several diseases and conditions have been associated with taste disorders and a decline in gustatory function is very common in the elderly.

The flavor test was previously developed, validated and patented by our group. It consists of a series of 20 aromatic extracts, corresponding to routine dietary use flavors for Italian people.

Each tastant, originally stored in a 30 mL amber bottle, is diluted in distilled water and stored at 4 °C, then it is kept at room temperature for 20 min before administration.

An aliquot of approximately 0,5 mL of each tastant is administered in the oral cavity using a 3mL Transfer Pipet and left for approximately 5 seconds; the mouth is then rinsed twice with distilled water before the administration of the following tastant.

At each administration, participants are invited to identify the aromatic by making a choice from 5 proposed items. A total of 21 aromatics (including one blank) are administered sequentially. The flavor score (FS) is calculated as the sum of correctly identified aromatics and ranged from 0 to 21.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Exclusion Criteria:

Allergies, drug usage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General population volunteerly selected during a project to investigate the role of lifestyle in preventing chronic diseases supported by the Campus Salute association (www.campussalute.it).
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Flavor score | Immediately after the test administration flavor score was calculated
  A flavor score (1-21) was measured in all the studied subjects using the Flavor test

CONTACTS AND LOCATIONS:
Overall Officials: Paolo E. Macchia, M.D., Ph.D., Principal Investigator — Dipartimento Medicina Clinica e Chirurgia, Università degli Studi di Napoli Federico II

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maione L, Cantone E, Nettore IC, Cerbone G, De Brasi D, Maione N, Young J, Di Somma C, Sinisi AA, Iengo M, Macchia PE, Pivonello R, Colao A. Flavor perception test: evaluation in patients with Kallmann syndrome. Endocrine. 2016 May;52(2):236-43. doi: 10.1007/s12020-015-0690-y. Epub 2015 Jul 25. PMID 26209039
- [Derived] Nettore IC, Maione L, Palatucci G, Dolce P, Franchini F, Ungaro P, Belfiore A, Colao A, Macchia PE. Flavor identification inversely correlates with body mass index (BMI). Nutr Metab Cardiovasc Dis. 2020 Jul 24;30(8):1299-1305. doi: 10.1016/j.numecd.2020.04.005. Epub 2020 Apr 20. PMID 32513578